CLINICAL TRIAL: NCT00429455
Title: Survey of the Need for Information on Fertility and Menopause-Related Treatment Effects Among Young Women Who Underwent Hematopoietic Stem Cell Transplantation
Brief Title: Survey of the Need for Information on Fertility and Menopause-Related Treatment Effects Among HSCT Patients
Status: Completed | Type: Observational
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 2005-0997
Record Dates: First submitted 2007-01-29; First posted 2007-01-31 (Estimated); Last update posted 2012-08-01 (Estimated); Status verified 2012-07

CONDITIONS: Stem Cell Transplantation
Keywords: Fertility; Menopause; Hematopoietic Stem Cell Transplantation; Questionnaire; Survey
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Survey Participants: Female patients who had a hematopoietic stem cell transplantation between January 1987 and September 2004 at M. D. Anderson Cancer Center.
  Interventions: Behavioral: Survey

INTERVENTIONS:
Behavioral: Survey — 3-Part Questionnaire

SUMMARY:
Primary Objective:

- To understand the importance of receiving information on fertility- and menopause-related treatment effects for female patients undergoing hematopoietic stem cell transplantation.

DETAILED DESCRIPTION:
Researchers are currently conducting a survey on how important it is to women who are having a stem cell transplant to have information about the effects of the treatment on their fertility (their ability to have children) and on the risk of early menopause. Researchers know that some women who had transplants think that the information that they received may have been lacking or was not appropriate for their needs. Therefore, researchers would like to ask women who have had stem cell transplants at M. D. Anderson Cancer Center to report what kind of information they got and would like to have gotten before or during their treatment.

ELIGIBILITY:
Inclusion Criteria:

* Female patients who had a hematopoietic stem cell transplantation between January 1987 and September 2004 at M. D. Anderson Cancer Center.
* Age 16 to 50 years at the time of the transplant.

Exclusion Criteria:

* History of ovarian cancer.
* History of hysterectomy/oophorectomy
* Non-English speaking patients

Ages: 16 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Female patients who had a hematopoietic stem cell transplantation between January 1987 and September 2004 at M. D. Anderson Cancer Center.
Sampling Method: Probability Sample
Enrollment: 196 (Actual)
Dates: Start 2007-03; Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
Number of Survey Responders | 2 Years

CONTACTS AND LOCATIONS:
Overall Officials: Naoto Ueno, MD, PhD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- U.T. M.D. Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: UT MD Anderson Cancer Center — http://www.mdanderson.org